CLINICAL TRIAL: NCT04224818
Title: Dual Trigger in the Final Oocyte Maturation in Poor Ovarian Responders: A Prospective Randomized Controlled Trial
Brief Title: Dual Trigger in the Final Oocyte Maturation in Poor Ovarian Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2018-0020
Record Dates: First submitted 2019-09-20; First posted 2020-01-13 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-01

CONDITIONS: Poor Ovarian Reserve
MeSH Terms: interventions — Triptorelin Pamoate; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual trigger (Experimental): Dual trigger: (0.3 mg GnRHa = triptorelin) with + HCG (Choriomon)10 000 IU . will be administered subcutaneously in a single dose 0.3 mg with 10 000 HCG when at least 2 follicles 18 mm in diameter have been observed by ultrasound examination.
  Interventions: Drug: Dual trigger
- hCG (standard) (Active Comparator): HCG (Choriomon) of 10 000 IU will be administered subcutaneously in a single dose when at least 2 follicles 18 mm in diameter have been observed by ultrasound examination.
  Interventions: Drug: hCG (standard)

INTERVENTIONS:
Drug: Dual trigger — Dual trigger: human Chorionic Gonadotropin (Choriomon 10,000 IU subcutaneous once) + Gonadotropin-Releasing Hormone agonist (Triptorelin 0.3 mg subcutaneous once)
  Other Names: Dual ovulation trigger (Choriomon and Triptorelin)
  Arms: Dual trigger
Drug: hCG (standard) — human Chorionic Gonadotropin (Choriomon 10,000 IU subcutaneous once)
  Other Names: human Chorionic Gonadotropin
  Arms: hCG (standard)

SUMMARY:
This is a randomized controlled clinical trial to investigate the effect of dual trigger (hCG and GnRH agonist) on the final oocyte maturation compared to the standard hCG trigger in patients with poor ovarian reserve seeking IVF/ICSI treatment.

DETAILED DESCRIPTION:
Women with POR (Bologna criteria) manifest a very low follicular response to controlled ovarian stimulation irrespective of the stimulation protocol utilized. Dual triggering of oocyte maturation was shown to improve follicle collection yield and oocyte maturation in women with predicted normal ovarian response. These benefits have been attributed to the GnRHa-induced FSH surge believed to promote oocyte nuclear maturation and cumulus expansion. The aim of the study is to show whether the co-administration of a GnRH agonist and hCG for final oocyte maturation improve oocyte collection and maturation rate

ELIGIBILITY:
Inclusion Criteria:

* Normal uterine cavity (as assessed by hysteroscopy or HSG).
* Normal hormonal investigation: TSH, PRL.
* Low ovarian reserve patients (AMH<1.5ng/ml, AFC of 7 or less, 5 oocytes or less retrieved in a previous cycle)

Exclusion Criteria:

* Abnormal uterine cavity (Hysteroscopy or HSG)
* Evidence of untreated endocrine disorders (abnormal TSH, prolactin, testosterone and androstenedione concentrations)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved (oocyte collection rate) | 38 hrs
  the total number of oocytes retrieved divided by the number of follicles aspirated (diameter ≥10 mm) on the day of oocyte retrieval
Number of mature oocytes (oocyte maturation rate) | 38 hrs
  the ratio of MII oocytes to the number of collected oocytes

SECONDARY OUTCOMES:
Fertilization rate | 48 hrs
  the ratio of normal fertilized oocytes (2PN) to the number of oocytes used for fertilization
Clinical pregnancy rate | 7 weeks
  the presence of fetal cardiac activity confirmed by transvaginal ultrasound 7 weeks after embryo transfer
Implantation rate | 7 weeks
  the number of gestational sacs visualized on ultrasound examination divided by the number of embryos transferred
Miscarriage rate | 12 weeks
  the spontaneous loss of a clinical pregnancy occurring before 12 completed weeks of gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Ghina S Ghazeeri, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon